CLINICAL TRIAL: NCT06761404
Title: Non-invasive VNS in Stroke Recovery
Acronym: NOVIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Timea Hodics, Director, Interventional Neuro-Recovery Program, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00038365
Record Dates: First submitted 2024-12-13; First posted 2025-01-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: taVNS; trans-auricular; non-invasive vagus nerve stimulation; stroke recovery; neuromodulation; rehabilitation; chronic stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Sham stimulation vs taVNS
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Sham Stimulation (Sham Comparator): Same procedure as with the active stimulation using the device's sham settings to elicit the same cutaneous sensation as the other stimulation conditions..
  Interventions: Device: taVNS
- taVNS (Experimental): Weak current (up to 0.8-4 mA) will be delivered using pulses according to standard protocol during each motor task for up to 90-minutes through surface electrodes which will be administered using the intensity identified as resulting in well tolerated skin sensation and best motor performance during our initial testing session.
  Interventions: Device: taVNS

INTERVENTIONS:
Device: taVNS — Experimental. The current will be increased gradually for both sham and real stimulation at the beginning of the 90-minute stimulation to lessen the itchy/numb skin sensation and to create the same skin sensation for subject blinding.

SUMMARY:
To evaluate feasibility and effectiveness of non-invasive VNS to enhance stroke recovery

DETAILED DESCRIPTION:
In this study, (Aim 1) we will test whether our non-invasive trans-auricular vagus nerve stimulation (taVNS) during occupational therapy task performance has the potential for large scale application through superior clinical benefit compared to sham in a broad group of stroke survivors including hemorrhagic strokes.

To determine the predictors of effective brain rewiring in the individual stroke patient, we will use an EEG and/or functional MRI (fMRI) connectivity biomarker independently of the success of the stimulation paradigm (Aim 2). We will test the hypothesis that better motor function will be associated with increased motor network connectivity pattern.

The central objective of this application is to determine whether taVNS significantly improves motor recovery for both ischemic and hemorrhagic strokes through increased connectivity as measured by a biomarker of plasticity. We address our objective through the following aims:

Aim 1: To determine the extent to which taVNS with concurrent occupational therapy (OT), causes significant, lasting motor gains in chronic stroke population

Hypothesis A: More chronic stroke patients treated with taVNS+OT will show clinically meaningful improved hand motor function over Sham+OT immediately after treatment as measured by upper extremity Fugl-Meyer (uFM) test response rate. 60 patients at least 6 months after ischemic or hemorrhagic stroke with persistent arm weakness will be enrolled in a 6-week double masked, sham-controlled, balanced parallel group design phase 2 clinical trial.

Hypothesis B: The sham group will achieve the same degree of motor function improvement in the open label cross-over phase as the original active taVNS group sustained clinical improvement after OT+VNS.

Hypothesis C: The open label home extension taVNS+OT phase will produce additional motor function improvement and will be associated with improved patient and caregiver satisfaction.

Aim 2: To determine the induced connectivity pattern of the brain resulting in the improved motor performance

Hypothesis A: Chronic stroke patients with improved motor performance will demonstrate increased connectivity between motor cortical areas as measured by high-definition EEG and/or fMRI functional connectivity compared to the non-responders immediately after treatment.

Hypothesis B: Network activation with taVNS is dependent on timing compared to movement and stimulation intensity. We will perform fMRI and /or high-definition EEG to evaluate network activity during taVNS at different intensity and phase of the movement.

This study evaluates the feasibility, efficacy and underlying plasticity changes of adjuvant noninvasive VNS to enhance motor recovery following ischemic and hemorrhagic strokes.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic ischemic or hemorrhagic stroke verified by computerized axial tomography or magnetic resonance imaging resulting in hemiparesis (MRC 1-4).
* Age more than 18, Male or Female, All racial and ethnic groups
* Entry into the study >6 months post onset
* Patients who can safely undergo taVNS
* Able to follow 2 step commands
* Modified Ashworth Scale Score =<3 in the involved upper extremity
* Passive range of motion within functional ranges at the shoulder, elbow, wrist and hand
* UFM =< 60 (scale 0-66)

Exclusion Criteria:

* Patients with history of severe alcohol or drug abuse, psychiatric illnesses like severe depression, poor motivational capacity, or severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as unable to follow study instructions).
* Patients with bilateral paresis, or weakness or sensory damage due to peripheral causes (e.g. peripheral nerve injury, muscle or orthopedic injury etc.)
* Subjects with contraindication to MRI of the brain
* Patients with severe uncontrolled medical problems (e.g. cardiovascular disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, or a deteriorated condition due to age, epilepsy or others).
* Patients with unstable cardiac arrhythmia, reentry tachycardia.
* Pregnancy
* Patients with pacemakers or stimulators that interfere with the stimulation, or other investigational devices or drugs
* Non-English speaking individuals will only be eligible if they can provide the appropriate translator for all the sessions of the study as no funding is available to pay for such services. However we plan to include them once funding has been secured in the subsequent larger trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate feasibility and effectiveness of non-invasive VNS to enhance stroke recovery | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]
  To determine the extent to which taVNS with concurrent occupational therapy (OT), causes significant, lasting motor gains in chronic stroke population
  Upper extremity Fugl-Meyer (uFM) The uFM test measures both proximal and distal upper extremity movements, ranges 0-66, higher score is better.

SECONDARY OUTCOMES:
To evaluate the biomarkers of plasticity associated with VNS | [Time Frame: Baseline 1(week 1), post-intervention (week 6), post intervention for sham crossover only (week 12)]
  We will use an EEG and/or functional MRI (fMRI) connectivity biomarker.
Wolf Motor Function Test (WMFT) | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]
  The WMFT is a time-based method to evaluate upper extremity performance while providing insight into joint-specific and total limb movements. This measurement includes video recording of the task performance where de-identifying will be attempted to the degree possible (face not in the frame, removing/blocking out identifying jewelry etc.). All patients will sign an informed consent explicitly authorizing such video-recording.
Functional upper extremity levels (FUEL) | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]
  The FUEL is an upper extremity post-stroke motor function classification system that does not require significant extra time or evaluator training.
NIH STROKE SCALE (NIHSS) | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]. Max score 42, minimum score 0. Score of 0 is best outcome
  The NIHSS is a standardized clinical examination to evaluate clinical functional impairment after stroke.
MRC grading scale | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]. Minimum score 0, max score 5 per item. 5 is normal, 0 is no movement.
  The MRC grading scale is a clinical scale to evaluate the motor impairment.
Timed up and Go | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]
  This test assesses gait speed, mobility, balance, walking ability and fall risk in older adults.
Barthel Index (BI) | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]. Minimum score 0, maximum score 100. Higher score is better
  The Barthel Index is an index measuring the patients' activities of daily living and of patient's independence in mobility and personal care.
Stroke Impact Scale (SIS) | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]. Minimum score 0, maximum score 100. 0 means no recovery, 100 means fully recovered
  A self-report questionnaire that evaluates disability and health-related quality of life after stroke from the perspective of the patient.
Zarit Burden Interview: Short (12-items) | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]
  Caregiver perspective questionnaire to assess caregiver burden. Additional caregiver questionnaire for perception of user friendliness, time savings, helpfulness, ease of use, perceived improvement and free comments will be collected.
Modified Rankin Scale (mRS) | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]
  Clinician-reported measure of global disability that has been widely applied for evaluating recovery from stroke and as a primary end point in randomized clinical trials (RCTs) of emerging acute stroke treatments.
Modified Ashworth Spasticity Scale | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]
  The modified Ashworth spasticity scale provides a rating of the degree of spasticity of a limb evaluated by clinical neurologic examination.
Quick Inventory of Depressive Symptomatology, Self-report (QIDS-SR) | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]. Minimum score 0, maximum score greater than 21. 0-5 means normal, greater than 21 is not
  A validated 16-item0-27 scale self-report questionnaire of depression.
taVNS questionnaire | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]
  Visual Analog Scale to prospectively evaluate taVNS effects such as skin sensation, tingling, skin redness etc. This will serve as a safety and tolerability measure.
Motor Activity log | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]
  A structured interview to assess how stroke survivors use their affected arm outside of the laboratory.
Wrist flexion-extension measurement | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]
  This measurement will be performed with our hand device to record maximum force of flexion and extension in standard arm position. taVNS test improvement will be calculated based on the speed and accuracy of the writs flexion measurement as described in our prior published work.
To determine the taVNS induced connectivity pattern of the brain | [Time Frame: Baseline, post intervention (week 6), post intervention (week 12), and follow up for the sham crossover group (week 18)]
  Primary outcome measure: Hypothesis A and Hypothesis B: Connectivity measure between motor cortical areas as measured by high definition EEG and fMRI functional connectivity in taVNS compared to Sham+OT immediately after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Timea Hodics, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States